CLINICAL TRIAL: NCT05390658
Title: Clinical Features and Risk Factors Analysis for Acute Myocardial Infarction Patients Received ECMO
Brief Title: Risk Factors Analysis for Acute Myocardial Infarction Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genglong Liu (Other)
Responsible Party: Sponsor-Investigator, Genglong Liu, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: ECOM
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: AMI - Acute Mesenteric Ischemia; Extracorporeal Membrane Oxygenation Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survival
  Interventions: Other: Not application
- Death
  Interventions: Other: Not application

INTERVENTIONS:
Other: Not application — Not application

SUMMARY:
ECMO has been used to save the lives of many critically ill patients with cardiorespiratory dysfunction as important rescue therapy. Though the proportion of ECMO applied to this population has been increasing year by year, clinical outcomes of AMI remain poor with high in-hospital mortality. Thus, it is necessary to characterize clinical features and investigate potentially modifiable factors contributing to outcomes of AMI patients who received ECMO treatment.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Alzheimer's Disease Age more than 18

Exclusion Criteria:

Life expectancy <1 year Prolonged cardiac arrest before VA-ECMO therapy (>60 min) Iatrogenic myocardial infarction secondary to a percutaneous coronary intervention VA-ECMO implanted in another center before admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: I. Clinical symptoms: the typical angina pectoris symptoms of acute myocardial infarction are compressive pain in the precardiac area and the back of the sternum, accompanied by sweating, a sense of dying, and a sense of suffocation. Taking nitroglycerin tablets or quick-effect Xusuxin pills cannot alleviate the symptoms.
  2. Typical ECG manifestations, such as pathological Q wave, ST-segment elevation, or pathological ST-segment depression, have corresponding lead changes.
  3. Increased myocardial enzymes, including CK, CK-MB, and troponin, etc. The diagnosis of acute myocardial infarction can be made with two of these three indicators.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2022-11-12 (Estimated); Study Completion 2023-01-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 1 month
  Survival information from ICU entry to ICU exit

CONTACTS AND LOCATIONS:
Locations (1):
- Genglong Liu, Guangzhou, State..., China

IPD SHARING:
Plan to Share IPD: Undecided